CLINICAL TRIAL: NCT04990401
Title: Adapted Tele-Behavioral Activation Targeted to Increase Physical Activity in Depression
Brief Title: Behavioral Activation Teletherapy to Increase Physical Activity
Acronym: BAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Madhukar H. Trivedi, MD, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2021-0441; 1R34MH122640-01A1 (NIH)
Record Dates: First submitted 2021-07-21; First posted 2021-08-04 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Depression; Depressive Disorder; Depressive Symptoms; Depressive Episode
Keywords: Therapy; Teletherapy; Physical Activity; Exercise
MeSH Terms: conditions — Depression; Depressive Disorder; Motor Activity

STUDY DESIGN:
Intervention Model Description: All eligible participants will receive the behavioral activation teletherapy intervention in this single-arm study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral Activation Teletherapy (Experimental): All eligible participants will be assigned to receive the behavioral activation teletherapy intervention.
  Interventions: Behavioral: Behavioral Activation Teletherapy

INTERVENTIONS:
Behavioral: Behavioral Activation Teletherapy — A total of 10 teletherapy sessions to be delivered over 12-14 weeks, designed to increase physical activity among depressed individuals.

SUMMARY:
This is a pilot study of acceptability, feasibility, and preliminary efficacy of a brief, 10-session Behavioral Activation intervention delivered via teletherapy to increase physical activity and treat depressive symptoms.

DETAILED DESCRIPTION:
This is a one-site, two-phase study that will use an initial group of individuals between the ages of 18 and 64 who have moderate to severe depressive symptoms and exercise less than 90 minutes a week. In both phases, participants will complete a total of 8 behavioral activation teletherapy sessions used to increase physical activity, followed by two biweekly booster sessions, for a total of 10 sessions. Participants will also complete weekly assessments remotely for both phases of the study. The screening visit and final intervention session will be in-person, and all other visits will be via telehealth. Participants will have the option to come to the clinic if they prefer.

In the initial phase (n = 15), participants who completed the intervention will have the option to participate in a focus group, and participants who partially completed the intervention will have the option to participate in a semi-structured interview. The total duration of phase one is 14 weeks. This initial phase will allow the researchers to refine and optimize the intervention to be delivered in the second phase.

In the second/pilot phase (n = 50), participants will complete a one-month and a two-month follow-up after the 10 intervention sessions. The total duration for phase two is 22 weeks.

Participants for both phases of the study will wear a Fitbit during the duration of their study participation, in order to record step count.

ELIGIBILITY:
Inclusion Criteria:

* Be18-64 years old;
* Able and willing to provide informed consent;
* Have moderate-to-severe depressive symptoms, with a PHQ-9 score ≥ 10;
* Insufficient moderate-to-vigorous physical activity (< 90 minutes a week);
* Demonstrated interest in increasing physical activity;
* Have a smartphone.

Exclusion Criteria:

* Have any current, past, or lifetime manic or hypomanic episode, psychosis, schizophrenia or schizophreniform disorder;
* Be currently experiencing active suicidal ideation (i.e. with suicidal thoughts, plan, and intent) or at a high risk for suicide during the course of the study, as designated by the PI;
* Have a medical condition that prohibits physical activity; be medically prohibited to exercise by primary care physician (PCP), OB-GYN (obstetrician-gynecologist) or study MD.
* Be in current, active psychotherapy

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Feasibility and acceptability - Screening | 1 week
  Number of participants screened per week (Goal 1-2 per week)
Feasibility and acceptability - Recruitment | 1 week
  Percentage of screened participants enrolled (Goal: 50%)
Intervention Adherence | Up to 14 weeks
  Percentage of intervention sessions attended (goal 75%)
Intervention Validity via Quality of Behavioral Activation Short Form | Up to 14 weeks
  Fidelity on supervisor's structured feedback form with average item score ≥3. The 14-item scale has each item ranging from 0-6, with higher values indicating higher levels of fidelity.
Participant retention | Up to 22 weeks
  Percentage of PHQ-9 assessments completed (Goal: 80%)
Participant outcome completion | Up to 22 weeks
  Percentage of valid Fitbit wear days > 12 hours (Goal: 80%)

SECONDARY OUTCOMES:
Depressive symptoms - 9-item Patient Health Questionnaire | Up to 22 weeks
  Change in self-Reported Depressive Symptoms, analyzed using linear mixed effects modeling controlling for baseline depressive symptoms and additional covariates
Physical activity - self-report days per week | Up to 22 weeks
  Change in self-reported frequency of physical activity (days per week), analyzed using linear mixed effects modeling controlling for baseline physical activity and additional covariates
Physical activity - self-report minutes per day | Up to 22 weeks
  Change in self-reported frequency of physical activity (minutes per day), analyzed using linear mixed effects modeling controlling for baseline physical activity and additional covariates
Physical activity - Fitbit step counter active minutes | Up to 22 weeks
  Change in objective data from Fitbit of "active minutes", using linear mixed effects modeling controlling for baseline physical activity and additional covariates
Physical activity - Fitbit step counter step count | Up to 22 weeks
  Change in objective data from Fitbit of "step count", using linear mixed effects modeling controlling for baseline physical activity and additional covariates

OTHER OUTCOMES:
Mediation of intervention through a number of pathways | Up to 22 weeks, using mediating timepoints post-session at Weeks 0, 3 and 7
  Testing whether the physical activity to depression reduction pathway is mediated by changes in (a) positive and negative affect; (b) anhedonia, (c), fatigue, (d) self-esteem, (e) overall depressive symptoms and (f) emotion regulation. For each potential mediator, both a direct and indirect pathway will be tested. First, the mediational model should meet the goodness of fit criteria (e.g., a non-significant X2, fit indices greater than .90 and significant path coefficients) and second, when a direct effect path is added to the model this path is either non-significant or adds little improvement in the overall predictive value of the model (i.e., increase in R2).
Minimum number of therapy sessions needed to achieve depression remission | Up to 14 weeks
  The minimum number of completed therapy sessions (1-10) needed to achieve depression remission, analyzed through discrete-time survival analysis.
Depressive symptoms - IDS-SR | Up to 22 weeks
  Change in self-reported Inventory of Depressive Symptoms (IDS-SR), analyzed using linear mixed effects modeling controlling for baseline depressive symptoms and additional covariates

CONTACTS AND LOCATIONS:
Overall Officials: Chad Rethorst, PhD, Principal Investigator — University of Texas Southwestern Medical Center; Madhukar Trivedi, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
If other investigators are interested in accessing data, they may contact the principal investigator in writing.

REFERENCES:
- [Derived] Rethorst CD, Trombello JM, Chen PM, Carmody TJ, Goodman LC, Lazalde A, Trivedi MH. Pilot evaluation on an adapted tele-behavioral activation to increase physical activity in persons with depression: a single-arm pilot study. BMC Psychol. 2024 Nov 9;12(1):643. doi: 10.1186/s40359-024-02053-5. PMID 39522018

DOCUMENTS (1):
  • Informed Consent Form: English Informed Consent Form (2023-06-29): https://cdn.clinicaltrials.gov/large-docs/01/NCT04990401/ICF_000.pdf